CLINICAL TRIAL: NCT02269176
Title: 12 Week, Multi-center, Randomized, Double-blind, Double Dummy, Parallel Group Trial Comparing the Efficacy and Safety of 40 & 80 mg Telmisartan and 50 & 100 mg Losartan in the Treatment of 150 Pairs of Primary Hypertension Patients
Brief Title: Efficacy and Safety of Telmisartan and Losartan in Primary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.365
Record Dates: First submitted 2014-10-20; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Losartan

ARMS (2):
- Telmisartan (Experimental): Low dose of telmisartan, uptitrated to high dose in case no sufficient effect is observered
  Interventions: Drug: Low dose of telmisartan; Drug: High dose of telmisartan
- Losartan (Active Comparator): Low dose of losartan, uptitrated to high dose in case no sufficient effect is observered
  Interventions: Drug: Low dose of losartan; Drug: High dose of losartan

INTERVENTIONS:
Drug: Low dose of telmisartan
  Arms: Telmisartan
Drug: High dose of telmisartan
  Arms: Telmisartan
Drug: Low dose of losartan
  Arms: Losartan
Drug: High dose of losartan
  Arms: Losartan

SUMMARY:
Using Losartan as a comparator, to evaluate the efficacy and safety of telmisartan in the treatment of the mild to moderate primary hypertension patients in China

ELIGIBILITY:
Inclusion Criteria:

- Mild to moderate primary hypertension, the mean sitting valley value of diastolic blood pressure (DBP) ≥ 95 and < 110 mmHg, and the mean sitting valley value of systolic blood pressure (SBP) < 180 mmHg

Exclusion Criteria:

- Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2000-07; Primary Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Changes in mean sitting valley value of DBP | 8 weeks after start of treatment
  The valley value of blood pressure refers to the blood pressure measured prior to the next administration of antihypertensives